CLINICAL TRIAL: NCT07012239
Title: The Frequency of Thiopurine Methyltransferase Polymorphism in Systemic Lupus Erythematosus Patients and Its Association With Azathioprine-Induced Adverse Effects
Brief Title: The Frequency of Thiopurine Methyltransferase Polymorphism in Systemic Lupus Erythematosus SLE
Acronym: TPMT
Status: Completed | Type: Observational
Sponsor: Bangladesh Medical University (Other)
Responsible Party: Principal Investigator, Mohammad Abul Kalam Azad, Associate Professor, Bangladesh Medical University
Other Study IDs: BSMMU/2016
Record Dates: First submitted 2025-05-31; First posted 2025-06-10 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-05

CONDITIONS: Genetic Polymorphism
Keywords: Azathioprine ,TPMT, Systemic lupus Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — Azathioprine

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- TPMT: TPMT positive in Azathioprine treated adverse effect positive
  Interventions: Drug: Azathioprine (AZA); Drug: TPMT

INTERVENTIONS:
Drug: Azathioprine (AZA) — Patient fulfilled indication of AZA Maintenance of remission of lupus nephritis, Neuro-psychiatric lupus, vasculitis, intolerance to steroid, associate with Defuse Parenchymal Lung Disease (DPLD) Starting AZA at a dose of 1 mg/kg/ body weight
  First follow-up at 2nd week and change dose of AZA 2 mg /kg/ BW/day
  Then Follow-up 4 weekly for total 12 week
  Not adverse effect of Azathioprine
  Other Names: Adverse effect of Azathioprine in SLE
Drug: TPMT — Adverse effect of azathioprine in SLE

SUMMARY:
ABSTRACT Background: Thiopurine S-methyltransferase (TPMT) is the rate-limiting enzyme for azathioprine (AZA) metabolism. Polymorphisms of this gene induce adverse effects of AZA. AZA is widely used as an immunosuppressant agent for the remission maintenance of Systemic Lupus Erythematosus (SLE). Objective: To study the frequency of TPMT polymorphism in SLE patients. Methods and Materials: This observational nested case control study was conducted in the department of Rheumatology (BMU) and Pharmacokinetics and Pharmacogenetics Laboratory, department of Pharmacy, Dhaka University (DU), Dhaka, from July 2014 to January 2016. 348 (aged 18-65 years) SLE patients were enrolled, 11 were excluded, and 337 were included. Among them, 120 patients took AZA. All patients gave informed written consent. We included the patient who fulfilled ACR criteria for SLE and excluded the following patients: pregnant woman, taking another myelosuppressive or experimental drug, recent blood transfusion, and unwilling patient. A five ml blood sample was collected from each patient and analyzed for a genetic study. The polymerase chain reaction-restriction fragment length polymorphism (PCR-RFLP) technique was used to detect the gene. The individual patient's disease activity was evaluated using the Systemic Lupus Erythematosus Disease Activity Index (SLEDAI). The chi-square test was used to compare the frequency of alleles in SEE patients who received AZA. Results: A total of 348 SLE patients accepted the request to participate. DNA was not isolated from 11 patients, and they were excluded from this study. The remaining 337 patients were evaluated. The patients were divided into two groups: one was the AZA group and the other was the non-AZA group. In the AZA group, there were 120 patients, and in the non-AZA group, there were 217 patients. Nine patients of the AZA group were not included, and they were recorded as drop-out patients because they did not complete the follow-up visits. Mean age in the AZA group was 28.41±9.5 years and in the non-AZA group27.27±8.6 years. Mean weight in the AZA group was 53.2±6.5 kg, and in the non-AZA group was 53.01±6.8. Male patients were 13 (3.35%), and female patients were 324 (96.65%). In this study 12 patients TPMT polymorphism and the frequency was 3.56%. Among the 12 polymorphism patients a had TPMT3C mutant allele. There was no TPMT3A and TPMT2 mutant alleles found this study population. Total 10 patients developed myelosuppression. Among them (60%) had TPMT polymorphism and 4 (40%) had no TPMT polymorphism. In AZA group 7 patients had TPMT polymorphism, 6 (85.7%) patients developed myelosuppression and 1 (14.3%) patient did not develop it (myelosuppression). In AZA group was 53.2±6.5 kg and in non-AZA group was 53.01±6.3. Male patients were 13 (3.35%) and female patients were 324 (96.65%). In this study 12 patients TPMT polymorphism and the frequency was 3.56%. Among the 12 polymorphism patients all had TPMT3C mutant allele. There was no TPMT3A and TPMT2 mutant alleles found in this study population. Total 10 patients developed myelosuppression. Among them 6 (60%) had TPMT polymorphism and 4 (40%) had no TPMT polymorphism. In AZA group 7 patients had TPMT polymorphism, 6 (85.7%) patients developed myelosuppression and I (14.3%) patient did not develop it (myelosuppression). In myelosuppressed patients all of them developed anaemia and leucopoenia. Seven of the 10 patients developed thrombocytopenia and pancytopenia. A total of 16 (14.44%) patients developed AZA-induced adverse effects (including myelosuppression). Two patients developed hepatotoxicity who had TPMT genetic polymorphism, but the rest of the nonhematological adverse effects developed in patients without the genetic polymorphism.

Conclusion: The frequency of TPMT polymorphism in this series of Bangladeshi SLE patients is 3.56%. Most of the patients with TPMT gene polymorphism developed AZA-induced myelosuppression. The hematological adverse effects of AZA were present both in patients with and without the genetic polymorphism

DETAILED DESCRIPTION:
In this study, we observed adverse effects, TPMT polymorphism, and disease status.

Objective: Primary- to observe the frequency of thiopurine methyltransferase (TPMT) polymorphism and its effect on the use of AZA in SLE. Secondary - to determine the frequency of TPMT polymorphism in SLE with or without AZA-induced adverse effects, and to determine the frequency of adverse effects of AZA in SLE patients.

Methods and Materials: This observational nested case-control study was done in the Department of Rheumatology at Bangladesh Medical University and the Pharmacokinetics and Pharmacogenetics laboratory in the Department of Pharmacy at Dhaka University. The study period was July 2014 to January 2016. A total of 330 people were included in this study. The study population was SLE patients attending lupus clinics and inpatient clinics. A Convenient sampling procedure was used.

After receiving informed consent from the patient, those who fulfilled the updated 1997 revised ACR criteria of SLE were included in this study. The patient was unwilling to participate, had received a recent blood transfusion, had been administered any other myelosuppression drug, and had received treatment interfering with the metabolism of AZA or 6 MP, like allopurinol or diuretics. Concomitant treatment with cyclosporine, Mycophenolate Mofetil, and pregnancy were excluded from the study.

Flow chart of study procedure: Part A IRB Clearance

SLE patient (Fulfilling 1997 ACR Criteria)

Blood sample collection

Isolation of Lymphocyte

DNA isolation from lymphocyte

PCR and Identification of TPMT Gene

Part B:

Patient fulfilled indication of AZA Maintenance of remission of lupus nephritis, Neuro-psychiatric lupus, vasculitis, intolerance to steroid, associate with Defuse Parenchymal Lung Disease (DPLD) Starting AZA at a dose of 1 mg/kg/ body weight

First follow-up at 2nd week and change dose of AZA 2 mg /kg/ BW/day

Then Follow-up 4 weekly for total 12 week

Quality assurance strategy All the patients were selected very carefully from the SLE clinic and the inpatient department of BSMMU under the supervisor's guidance. The patients who were able to give their complete history will be interviewed only; those who were mentally unstable, very ill to give their history, or who lost their medical document will be excluded from the study. Information gathered from the patient was checked and rechecked with the medical record. To ensure the drug ingestion, we asked each patient to show the empty drug strip in every visit. Data collection per the questionnaire was scrutinized for quality assurance of interviewing and to check the standardization of the questionnaire. Any changes or corrections to the questionnaire and the data collection strategy were made per the guide's advice. A midterm evaluation of the study was done to check the consistency of data collection. In case of any incomplete data, we interviewed the patient again to get all the required information. Data cleaning was done before editing on the computer for analysis.

Ethical issues The nature and purpose of the study were explained in detail to all participants. The relevant investigation was done, and treatment was given to all subjects in this study. Informed and written consent was taken from every patient before enrollment. A unique identification number was provided to each patient. Each patient enjoyed every right to participate, refuse, or withdraw from the study at any point, but proper treatment will be ensured even then. Before starting this study, ethical clearance was taken from the Institutional Review Board (IRB), BSMMU. Data taken from the patients was regarded as confidential and kept locked under the principal investigator for purposeful use only.

Analysis After collecting information, all data were checked, verified for consistency, and edited appropriately. Simple descriptive measures like percentage, mean, and standard deviation of different variables were calculated. Variables were described as mean and standard deviation for quantitative data. The chi-square test was used to compare the prevalence of polymorphism alleles in SLE patients who received and did not receive AZA. The Mann-Whitney test was used for nonparametric data. A Z test was used to compare the proportion. The difference between means was compared using the Mann-Whitney U test. A p-value less than or equal to 0.05 was considered significant. All data analysis was done using the SPSS/PC statistical software package.

ELIGIBILITY:
Inclusion Criteria:

* Who fulfilled the updated 1997 revised ACR criteria of SLE were included in this study

Exclusion Criteria:

The patient was unwilling to participate Had received a recent blood transfusion Had been administered any other myelosuppression drug Had received treatment interfering with the metabolism of AZA or 6 MP, like allopurinol or diuretics Concomitant treatment with cyclosporine, Mycophenolate Mofetil, and pregnancy were excluded from the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 330 people were included in this study. The study population was SLE patients attending lupus clinics and inpatient clinics. A Convenient sampling procedure was used
Sampling Method: Probability Sample
Enrollment: 348 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2017-01-01 (Actual); Study Completion 2018-01-01 (Actual)

PRIMARY OUTCOMES:
Adverse effect of azathioprine in SLE | 4 weekly for 12 week
  SLADAI Score in SLE

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad AK Azad, Principal Investigator — Associate professor
Locations (1):
- Mohammad Abul Kalam Azad, Dhaka, Bangladesh